CLINICAL TRIAL: NCT05907460
Title: EXecution of Trans-Esophagus Echo Cardiogram in CardioPulmonary Resuscitation for Patients With Out-of-hospital Cardiac Arrest
Acronym: EXECT_CPR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 109070-F
Record Dates: First submitted 2023-06-08; First posted 2023-06-18 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-02

CONDITIONS: Out-Of-Hospital Cardiac Arrest
Keywords: Out-Of-Hospital Cardiac Arrest; Chest compression site; transesophageal echocardiography; end-tidal CO2
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Masking Description: This is an open label study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Perform standard advanced life support. No examination of transesophageal echocardiography during cardiopulmonary resuscitation.
- Intervention group (Experimental): Perform examination of transesophageal echocardiography during cardiopulmonary resuscitation and adjust the chest compression site to avoid left ventricular outflow tract according to the result of transesophageal echocardiography
  Interventions: Device: transesophageal echocardiography examination during cardiopulmonary resuscitation

INTERVENTIONS:
Device: transesophageal echocardiography examination during cardiopulmonary resuscitation — Perform transesophageal echocardiography in patients with out-of-hospital cardiac arrest during cardiopulmonary resuscitation and adjust the chest compression site to compress the left ventricle and avoid left ventricular outflow tract.
  Arms: Intervention group

SUMMARY:
The purpose of this single center, randomized clinical control trial is to determine that changing chest compression site during cardiopulmonary resuscitation according to the examination of the TEE could increase the level of end-tidal CO2, which represents the quality of cardiopulmonary resuscitation, or not in adult patients with non-traumatic out-of-hospital cardiac arrest while comparing to those who don't receive examination of transesophageal echocardiography during cardiopulmonary resuscitation.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 20 years-old
2. Out-of-hospital cardiac arrest
3. Non-trauma

Exclusion Criteria:

1. Obvious signs of death appears, such as separation of head and body, rigor mortis, livor mortis, cankered corpse......etc.
2. Family members clearly express the willing of do not attempt resuscitation or patients who have registered advance care planning not to attempt resuscitation.
3. Patients not suitable for transesophageal ultrasound, such as patients with esophageal tumor, those whose probe cannot be placed......etc.
4. Received Extracorporeal CPR.
5. Achieving sustained ROSC before ED arrival

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2023-06-29 (Actual); Primary Completion 2023-11-19 (Actual); Study Completion 2023-11-19 (Actual)

PRIMARY OUTCOMES:
Rate of sustained return of spontaneous circulation (ROSC) | 20 minutes after ROSC
  successful restoration and maintenance of a patient's heartbeat and blood circulation after undergoing cardiopulmonary resuscitation (CPR) for at least 20 minutes

SECONDARY OUTCOMES:
Rate of any return of spontaneous circulation | 1 minutes after ROSC
  successful restoration and maintenance of a patient's heartbeat and blood circulation after undergoing cardiopulmonary resuscitation (CPR)
Rate of survival to ICU admission | 48 hours after ROSC
  Successful restoration and stabilization of a patient's heartbeat and circulation, enabling safe transfer to the ICU.
Rate of survival to discharge | 6 months after ROSC
  successful restoration and maintenance of a patient's heartbeat and blood circulation and able to complete treatment course till discharge
Rate of discharge with favorable neurological outcomes | 6 months after ROSC
  using cerebral performance category score to measure neurologic outcomes of the patient at the time while patient's discharge. CPC1 and 2 are consider as favorable neurological outcomes, CPC3 and 4 are consider as unfavorable neurological outcomes
end-tidal carbon dioxide (EtCO2) | During resuscitation
  measuring end-tidal carbon dioxide during resuscitation

CONTACTS AND LOCATIONS:
Overall Officials: Jun-Tang Sun, MD, Msc, Study Chair — Attending physician of emergency medicine department
Locations (1):
- Far Eastern Memorial Hospital, Banqiao District, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No